CLINICAL TRIAL: NCT06602466
Title: A 4-Week Randomised, Controlled, Examiner-blind, Clinical Study Investigating the Efficacy of an Experimental Toothpaste Containing Stannous Fluoride in Improving Gingival Health
Brief Title: A Clinical Study Investigating the Effect of an Experimental Toothpaste Containing Stannous Fluoride in Improving Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300178
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will brush their teeth with full ribbon of test toothpaste on head of toothbrush for one timed minute twice a day (morning and evening) for 4 weeks.
  Interventions: Drug: Test toothpaste
- Reference Toothpaste (Negative Control) (Active Comparator): Participants will brush their teeth with full ribbon of reference toothpaste (Colgate Cavity Protection) on head of toothbrush for one timed minute twice a day (morning and evening) for 4 weeks.
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Test toothpaste — 0.454% Stannous Fluoride, 0.3% Zinc Chloride,1% Alumina toothpaste containing 1100 parts per million (ppm) fluoride.
  Arms: Test Toothpaste
Drug: Colgate Cavity Protection Toothpaste — Commercial toothpaste containing 1450 ppm fluoride.
  Arms: Reference Toothpaste (Negative Control)

SUMMARY:
The aim of this 4-week clinical study is to evaluate the ability of an experimental toothpaste, containing 0.454 percent (%) Stannous Fluoride (SnF2), 0.3% Zinc Chloride (ZnCl2) and 1% Alumina, to improve gingival health and plaque accumulation compared to a regular fluoride toothpaste (negative control) in participants with plaque-induced mild to moderate gingivitis.

DETAILED DESCRIPTION:
This will be a single-center, 4 weeks, randomized, controlled, examiner-blind, 2 treatment arms, stratified, parallel group design clinical study, investigating gingival health and supra-gingival plaque reduction on healthy participants after using an experimental toothpaste containing 0.454% SnF2, 0.3% ZnCl2 and 1% Alumina. Sufficient participants will be screened so that at least 160 participants are randomized (approximately 80 per group) to ensure approximately 144 (approximately 72 per group) evaluable participants complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Biological sex at birth was male or female.
* Aged 18 to 70 years inclusive, at the signing of the informed consent.
* Willing and able to comply with scheduled visits, treatment plan, saliva sample collection, study restrictions, Lifestyle Considerations and other study procedures.
* In good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant oral health that meets all the following:

At Screening (Visit 1):

* Participant with at least 20 natural, permanent teeth, (excluding 3rd molars).
* Participant with at least 40 evaluable surfaces for MGI, BI, and TPI.
* A healthy participant with mild to moderate plaque-induced gingivitis in the opinion of the clinical examiner.
* Overall MGI less than or equal to (<=) 1.75 to <= 2.30

At Baseline (Visit 2):

* Overall MGI greater than or equal to (>=) 1.75 to <= 2.30
* Overall TPI score >= 1.5

Exclusion Criteria:

* An employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator (or medically qualified designee), an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (for example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study outcomes and/or participant safety.
* A participant who is pregnant (self-reported) or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to any study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who is a current smoker or an ex-smoker (including vaper) who stopped within 6 months of Screening.
* A participant who is using smokeless forms of tobacco (for example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding.
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (for example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* Medications exclusions: At Screening (Visit 1):

  1. A participant using any antibiotic medication within 28 days prior to screening or at any time during the study.
  2. Participant who has used an anti-bacterial toothpaste/mouthwash (for example, chlorhexidine) or another oral care product within 2 weeks of Screening that, in the opinion of the investigator or dentally qualified designee, could affect gingival health, plaque formation or oral bacteria.
  3. A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
  4. A participant currently taking a systemic medication (for example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers, statins).
* Medications exclusions: At Baseline (Visit 2):

  1. A participant who has taken any antibiotics during the washout period (between Screening and Baseline).
  2. A participant who has taken (in the previous 14 days) a systemic medication (for example, anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  3. A participant who has used an antibacterial dentifrice or mouthwash (for example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with gingival health, plaque formation and oral bacteria, in the period between Screening and the Baseline visit.
* Periodontal exclusions:

  1. A participant who shows signs of periodontitis [at both Screening (Visit 1) and Baseline visits (Visit 2)].
  2. A participant with a Basic Periodontal Examination (BPE) score of 4 or above in one or more sextants.
  3. A participant with BPE score >= 3, if with probing pocket, a single tooth dept is >= 5 mm.
  4. A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  5. A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
* Dental Exclusions:

  1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  2. A participant who has dentures (partial or full).
  3. A participant who has an orthodontic appliance (bands, appliances, or fixed/ removable retainers).
  4. A participant who received orthodontic therapy within 3 months of Screening.
  5. A participant who has numerous restorations in a poor state of repair.
  6. A participant who has any dental condition (for example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  7. A participant who has had dental prophylaxis within 12 weeks of Screening.
  8. A participant who has had teeth bleaching within 12 weeks of Screening.
  9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham University Dental School, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in United Kingdom.
Pre-assignment Details: A total 175 participants were enrolled; 161 participants were randomized to a treatment (80 participants in the test product group and 81 participants in the reference product group). Total 154 participants completed the study (76 participants in the test product group and 78 participants in the reference product group).
Groups:
- Test Toothpaste: Participants were instructed to brush their teeth with full ribbon of test toothpaste (containing 0.454 percent [%] Stannous Fluoride, 0.3% Zinc Chloride,1% Alumina) on head of toothbrush for one timed minute twice a day (morning and evening) for 4 weeks.
- Reference Toothpaste (Negative Control): Participants were instructed to brush their teeth with full ribbon of reference toothpaste (Colgate Cavity Protection) on head of toothbrush for one timed minute twice a day (morning and evening) for 4 weeks.
Period: Overall Study
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Started | 80 | 81
Completed | 76 | 78
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all randomized participants who received at least one dose of the investigational product. Post randomization, two participants (from test group) received incorrect study product (i.e. Reference product). The Safety Population is presented using actual study product received and thus, the Overall Number of Baseline Participants in "Reference Toothpaste (Negative Control)" is greater than the number of participants included in the Participant Flow module.
Groups:
- Test Toothpaste: Participants were instructed to brush their teeth with full ribbon of test toothpaste (containing 0.454% Stannous Fluoride, 0.3% Zinc Chloride,1% Alumina) on head of toothbrush for one timed minute twice a day (morning and evening) for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control) | Total
Number analyzed (Participants) | 78 | 83 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (11.75) | 27.9 (11.76) | 27.5 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 34 | 39 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 78 | 83 | 161
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 5 | 3 | 8
  Asian - Central/South Asian Heritage | 26 | 29 | 55
  Asian - East Asian Heritage | 4 | 6 | 10
  Asian - South East Asian Heritage | 6 | 6 | 12
  White - Arabic/North African Heritage | 3 | 7 | 10
  White - White/Caucasian/European Heritage | 29 | 28 | 57
  Multiple | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Bleeding Index (BI) at Week 4
Description: The BI is an invasive assessment of gingival bleeding performed using a round-end probe. Presence/absence of gingival bleeding was assessed for 30 seconds after probing. BI was assessed on 3-points scale ranging from 0 to 2, where 0= Absence of bleeding on probing, 1= Bleeding observed within 30 seconds of probing, 2= Bleeding observed immediately on probing. Mean BI was calculated by taking the average over all tooth sites assessed for a participant. Lower score indicated improvement in the symptoms. Adjusted mean value was derived using ANCOVA model.
Time Frame: Week 4
Population: Modified Intent-To-Treat (mITT) Population comprised of all randomized participants who received at least one dose of investigational product and completed at least one-post Baseline BI assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 76 | 78
score on a scale | 0.19 (0.013) | 0.21 (0.013)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p = 0.2992, ANCOVA; Adjusted Mean Difference = -0.02, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.018

2. Secondary Outcome: Adjusted Mean Number of Bleeding Sites (NBS) at Week 4
Description: The bleeding assessment was done using round-end probe. The number of bleeding sites for each participant= the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Adjusted mean value was derived using ANCOVA model.
Time Frame: Week 4
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 76 | 78
bleeding sites | 30.0 (1.96) | 32.5 (1.93)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p = 0.3612, ANCOVA; Adjusted Mean Difference = -2.5, 95% CI 2-sided [-7.9 to 2.9], Standard Error of Mean 2.75

3. Secondary Outcome: Adjusted Mean Modified Gingival Index (MGI) at Week 4
Description: The MGI is a non-invasive visual assessment of gingival inflammation. MGI was assessed for all evaluable surfaces, four sites per tooth and was scored on a 5-point scale ranging from 0 to 4, where 0= Absence of inflammation, 4= Severe inflammation. Lower score indicated improvement in the symptoms. Adjusted mean value was derived using ANCOVA model.
Time Frame: Week 4
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 76 | 78
score on a scale | 1.79 (0.011) | 1.83 (0.010)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p = 0.0117, ANCOVA; Adjusted Mean Difference = -0.04, 95% CI 2-sided [-0.07 to -0.01], Standard Error of Mean 0.015

4. Secondary Outcome: Adjusted Mean Overall Turesky Plaque Index (TPI) at Week 4
Description: The TPI is a non-invasive assessment of supra-gingival plaque accumulation. The plaque was disclosed using a plaque disclosing dye solution and the TPI was assessed using a 6-point scale ranging from 0 to 5, where 0= No plaque, 5= Plaque covering 2/3 or more of the crown of the tooth. Lower score indicated improvement in the symptoms. Adjusted mean value was derived using ANCOVA model.
Time Frame: Week 4
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 76 | 78
score on a scale | 2.64 (0.037) | 2.62 (0.036)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p = 0.7616, ANCOVA; Adjusted Mean Difference = 0.02, 95% CI 2-sided [-0.09 to 0.12], Standard Error of Mean 0.052

5. Secondary Outcome: Adjusted Mean Interproximal TPI at Week 4
Description: as for outcome 4
Time Frame: Week 4
Population: mITT Population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
Number analyzed (Participants) | 76 | 78
score on a scale | 3.03 (0.039) | 3.03 (0.038)
Statistical Analysis 1: Comparison: Test Toothpaste vs Reference Toothpaste (Negative Control); Test type: Superiority; p = 0.9321, ANCOVA; Adjusted Mean Difference = -0.00, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.055

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 69 days).
Description: Post randomization, two participants (from test group) received incorrect study product (i.e. Reference product). The Safety Population is presented using actual study product received and thus, the Overall Number of Baseline Participants in "Reference Toothpaste (Negative Control)" is greater than the number of participants included in the Participant Flow module.
Arm/Group | Test Toothpaste | Reference Toothpaste (Negative Control)
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/83
Other Adverse Events (participants affected / at risk) | 13/78 | 6/83
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Toothpaste (N=78) | Reference Toothpaste (Negative Control) (N=83)
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 4 | 2
HYPERAESTHESIA TEETH (Gastrointestinal disorders) | 2 | 1
ORAL DISCOMFORT (Gastrointestinal disorders) | 2 | 0
TONGUE ULCERATION (Gastrointestinal disorders) | 1 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT06602466/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT06602466/SAP_001.pdf